CLINICAL TRIAL: NCT01156402
Title: Culturally-Appropriate Childhood Obesity Prevention Program for Hispanic Families
Brief Title: Childhood Obesity Prevention Program for Hispanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meharry Medical College (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 030425PC062 03 (Meharry IRB)
Record Dates: First submitted 2010-06-14; First posted 2010-07-02 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Obesity
Keywords: Obesity; Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Oral Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Intervention: Obesity Prevention (Experimental)
  Interventions: Behavioral: Healthy Families-Childhood Obesity Prevention and Oral Health
- Alternative Intervention/control: Oral Health (Experimental)
  Interventions: Behavioral: Healthy Families-Childhood Obesity Prevention and Oral Health

INTERVENTIONS:
Behavioral: Healthy Families-Childhood Obesity Prevention and Oral Health — The active intervention was adapted from the We Can! parent intervention to be culturally-appropriate for Hispanic families of children ages 5-7. The tailored intervention is based on Social Cognitive Theory and Behavioral Choice Theory to provide parents and children with cognitive and behavioral skills to enable change in the target behaviors, and to encourage them to practice using these skills to strengthen their perceived competence in using these behaviors effectively.

SUMMARY:
The purpose of this study is to evaluate the efficacy of a culturally-appropriate childhood obesity intervention with Hispanic families. The program aims at preventing childhood obesity by targeting parents to address nutrition, physical activity, and sedentary behaviors in their children.

DETAILED DESCRIPTION:
Childhood obesity has been ranked as a critical public health threat in the U.S. due to the increasing prevalence of obesity among children over the past three decades. Childhood obesity poses both intermediate and long-term health risks, as well as considerable economic costs. While this epidemic affects all socioeconomic levels, certain racial/ethnic groups are disproportionately affected, including Hispanics.The long-term goal of the current research is to contribute to the reduction of racial/ethnic disparities in obesity and obesity-related outcomes among Hispanics by testing a childhood obesity prevention program that has been culturally tailored for the Hispanic population through a participatory process. This developmental community-based participatory research (CBPR) project is a collaborative community-academic partnership between Meharry Medical College (MMC), Tennessee State University-Center for Health Research (TSU-CHR), and a grassroots community-based organization called Progreso Community Center (PCC). The Childhood Obesity Study is designed to evaluate two programs for Hispanic children ages 5 to 7 and their parents. One program focuses on nutrition and physical activity (based on NIH's "We Can!" program), and a parallel program focuses on oral health (developed by TSU's Dental Hygiene Program). Upon enrollment in the Study, parents and children will respond to an initial interview involving body measurement and questionnaire. Families will be given physical activity monitor to be worn for 7 days and randomly assigned to one of two groups. The families assigned to the Nutrition and Physical Activity Program will attend eight (8) bi-weekly classes (one every two weeks for four months) dealing with nutrition and physical activity. In the Oral Health Program families will attend 4 monthly classes (once a month for four months). These sessions deal with ways to take care of children's teeth and oral health. In addition, these families will have the opportunity to sign up for a free dental cleaning and assessment at the Dental Hygiene Clinic at Tennessee State University.

ELIGIBILITY:
Inclusion Criteria:

Children:

* 5-7 year-old female or male of Hispanic origin (identified by parent)
* resident of Davidson County or adjacent counties
* ≥25th percentile of age- and sex-specific BMI (CDC growth charts) or one parent/caregiver with BMI ≥ 25 kg/m2
* More than one child may enroll per family

Parents:

* Hispanic origin (self-identified)
* Spanish speaker
* adult age 18 or older
* parent of at least one eligible child
* Only one parent per family may enroll as a study participant and respond to questionnaires

Exclusion Criteria:

Children:

* BMI ≥ 35 kg/m2
* Medical conditions affecting growth
* Conditions limiting participation in the interventions or measurements
* Taking medications affecting growth
* No consent or inability to understand informed consent
* Incomplete or missed baseline assessments
* Plan to move from geographic area within the next 12 months.

Parents:

* No exclusions

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 319 (Actual)
Dates: Start 2010-05; Primary Completion 2013-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI)-for-age percentile | one year

SECONDARY OUTCOMES:
Child eating behaviors | One year
Child physical activity (accelerometers) | One year
Parenting strategies | One year
parent physical activity | one year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Vanderbilt University, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee

REFERENCES:
- [Background] Zoorob R, Buchowski MS, Beech BM, Canedo JR, Chandrasekhar R, Akohoue S, Hull PC. Healthy families study: design of a childhood obesity prevention trial for Hispanic families. Contemp Clin Trials. 2013 Jul;35(2):108-21. doi: 10.1016/j.cct.2013.04.005. Epub 2013 Apr 26. PMID 23624172